CLINICAL TRIAL: NCT01035320
Title: Platelet Function in Diabetic Patients With and Without Renal Impairment, and the Effects of Lipid Lowering Treatment
Acronym: PLAUDIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Paul Hjemdahl, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2004-004416-22 DMK001
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus; Impaired Renal Function
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- simvastatin + ezetimibe (Experimental): Cross-over study with placebo only run-in period. All patients participate in this arm with simvastatin + ezetimibe either as first treatment period (8-10 weeks)or second treatment period (8-10 weeks). The primary comparison is ezetimibe vs. placebo on top of simvastatin. A secondary comparison will be simvastatin vs. placebo run-in.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — After a placebo only run-in period patients (two groups) are treated with simvastatin + ezetimibe and simvastatin + placebo in a cross-over trial. Ezetimibe effects on top of simvastatin will be evaluated as the primary aim; simvastatin effects compared to run-in on placebo will be evaluated as a secondary aim.
  Other Names: Simvastatin; Ezetrol

SUMMARY:
The purpose of this study is compare the effects of simvastatin+ezetimibe with those of simvastatin alone on platelet activity, platelet-leukocyte interactions and inflammatory variables in diabetic patients with or without impaired renal function.

DETAILED DESCRIPTION:
A detailed study protocol is available.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or type 2
* With or without established microalbuminuria (albumin-to-creatinine ratio (ACR)2,5-25 mg/mmol for men, and 3,5-25 mg/mmol for women, according to ISH and ESC recommended criteria)
* Glomerular filtration rate (GFR) between 15-60 ml/min/1.73m2 (measured the last 6 months) or GFR >75ml/min/1.73m2. The abbreviated Modification of Diet in Renal Disease (MDRD) equation will be used to calculate GFR.
* Age 18-80 years

Exclusion Criteria:

* Definite history of myocardial infarction, coronary revascularisation procedure or stroke. (i.e, a strong clinical indication for statin treatment)
* Functioning renal transplant, or living donor-related transplant planned.
* Patients on dialysis.
* Poor metabolic control, i.e HbA1c > 9%
* Definite history of chronic liver disease, or abnormal liver function (i.e ALT >1,5 x ULN or, if ALT not available, AST > 1,5 x ULN).
* Evidence of active inflammatory muscle disease (e.g dermatomyositis, polymyositis), or CK>3 x ULN;
* Definite previous adverse reaction to a statin or to ezetimibe
* Definite previous adverse reaction to acetylsalicylic acid.
* Definite previous adverse reaction to an ACE-inhibitor.
* Need for concomitant treatment with a strong inhibitor of CYP3A4, such as itrokonazole, ketokonazole, erythromycin, clarithromycin, HIV-protease inhibitors or nefazodone (i.e. agents that may markedly elevate simvastatin levels).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Compare the effects of simvastatin + ezetimibe with those of simvastatin alone, on thrombogenic mechanisms, in patients with diabetes mellitus type 2. | 6 weeks, 14-18 weeks, 22-24 weeks

SECONDARY OUTCOMES:
Compare effects of simvastatin alone with those of placebo on thrombogenic mechanisms. Compare the effects of simvast. + ezetim. with those of simvast. alone on inflammatory variables. Assess how the treatment effect relate to renal function. | 6 weeks, 14-18 weeks, 22-24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hjemdahl, MD, PhD, Principal Investigator — Dept. of Medicine, Clinical Pharmacology Unit, Karolinska University Hospital (Solna), Stockholm, Sweden
Locations (1):
- Department of Medicine, Clinical Pharmacology Unit, Karolinska University Hospital (Solna), Stockholm, Sweden

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Almquist T, Jacobson SH, Mobarrez F, Nasman P, Hjemdahl P. Lipid-lowering treatment and inflammatory mediators in diabetes and chronic kidney disease. Eur J Clin Invest. 2014;44(3):276-84. doi: 10.1111/eci.12230. Epub 2014 Jan 22. PMID 24720535
- [Derived] Almquist T, Jacobson SH, Lins PE, Farndale RW, Hjemdahl P. Effects of lipid-lowering treatment on platelet reactivity and platelet-leukocyte aggregation in diabetic patients without and with chronic kidney disease: a randomized trial. Nephrol Dial Transplant. 2012 Sep;27(9):3540-6. doi: 10.1093/ndt/gfs183. Epub 2012 Jun 13. PMID 22700717